CLINICAL TRIAL: NCT00104663
Title: PRION-1: Quinacrine for Human Prion Disease. A Partially Randomized Patient Preference Trial to Evaluate the Activity and Safety of Quinacrine in Human Prion Disease
Brief Title: PRION-1: Quinacrine for Human Prion Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.1; Grant ID:71361
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Prion Disease
Keywords: Creutzfeldt-Jakob disease; inherited; sporadic; acquired; new variant CJD
MeSH Terms: conditions — Prion Diseases; Creutzfeldt-Jakob Syndrome | interventions — Quinacrine

INTERVENTIONS:
Drug: Quinacrine

SUMMARY:
PRION-1 aims to assess the activity and safety of Quinacrine (Mepacrine hydrochloride) in human prion disease. It also aims to establish an appropriate framework for the clinical assessment of therapeutic options for human prion disease that can be refined or expanded in the future, as new agents become available.

DETAILED DESCRIPTION:
The human prion diseases have been traditionally classified into Creutzfeldt-Jakob disease (CJD), Gerstmann-Sträussler-Scheinker (GSS) disease and kuru. They can alternatively be classified into three causal categories: sporadic, acquired and inherited. The appearance of a new human prion disease, variant CJD (vCJD), in the United Kingdom from 1995 onwards, and the experimental evidence that this is caused by the same prion strain as that causing bovine spongiform encephalopathy (BSE) in cattle, has raised the possibility that a major epidemic of vCJD will occur in the United Kingdom and other countries as a result of dietary or other exposure to BSE prions. These concerns have led to intensified efforts to develop therapeutic interventions.

Quinacrine has been previously used to treat other diseases such as malaria; however, it was found to have serious side effects and is no longer licensed in the United Kingdom. There is only very limited evidence from laboratory tests for the potential use of quinacrine in human prion disease, and the evidence to date for any possible clinical benefit is very scarce. The PRION-1 trial is being undertaken since there are no other drugs currently available which are considered suitable for human evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years or more, diagnosed with any type of human prion disease.

Exclusion Criteria:

* In a coma, or in a pre-terminal phase of disease such that prolongation of the current quality of life would not be supported
* Known sensitivity to quinacrine
* Been taking any other putative anti-prion therapy for less than 8 weeks

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2004-06; Study Completion 2007-03

PRIMARY OUTCOMES:
Time to death
proportion of responders, with "responders" defined as patients showing either clinical improvement or lack of deterioration in 3 key neurological and neuropsychiatric measures

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE)
Clinician's Dementia rating (CDR)
Rankin score
Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Glasgow coma score
Barthel Activities of Daily Living (ADL)
magnetic resonance imaging scan (MRI)
electro-encephalogram (EEG)
cerebrospinal fluid (CSF)

CONTACTS AND LOCATIONS:
Overall Officials: John Collinge, MD, FRCP, Principal Investigator — MRC Prion Unit; Janet Darbyshire, MBChB, FRCP, Study Director — MRC Clinical Trials Unit
Locations (1):
- National Prion Clinic, London, United Kingdom

REFERENCES:
- See also: MRC Clinical Trials Unit — http://www.ctu.mrc.ac.uk/default.aspx?page=310